CLINICAL TRIAL: NCT06214013
Title: Proposal for an Adaptation of Linehan's Biosocial Model to Emotional Dysregulation in Autism Spectrum Disorder: Narrative Review of the Literature and Clinical Case
Brief Title: Adaptation of Linehan's Biosocial Model to Emotional Dysregulation in Autism Spectrum Disorder
Acronym: DE-TSA
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8726
Record Dates: First submitted 2023-12-14; First posted 2024-01-19 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2023-12

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Disorder
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Linehan's biosocial model conceptualizes the factors at play in the development of emotional dysregulation (ED), that is, difficulty regulating one's emotions, in borderline personality disorder (BPD). The model explains ED as the result of the interaction between the person's biological emotional vulnerability and their exposure to early invalidating experiences from those around them. Recently, ED has been shown to be prevalent in autism spectrum disorder (ASD). The objective of the study is to propose an adaptation of Linehan's model to the specificities of ASD to conceptualize the factors contributing to ED in the context of this disorder. To do this, the investigators will carry out a narrative literature review, as well as an illustrative case conceptualization based on the proposed model.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (≥18 years old)
* Having been diagnosed with ASD without intellectual disability
* Presenting severe ED with self-harming behaviors and/or suicidal behaviors

Exclusion Criteria:

- Subjects not meeting the study eligibility criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects (≥18 years old) Having been diagnosed with ASD without intellectual disability
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2023-02-21 (Actual); Primary Completion 2023-05-21 (Actual); Study Completion 2023-05-21 (Actual)

PRIMARY OUTCOMES:
Adaptation of Linehan's biosocial model to emotional dysregulation in autism spectrum disorder | The bibliography research will cover the period from 2015 to 2021.
  This study is based on a narrative literature review, and will propose an illustrative case conceptualization based on Linehan's biosocial model.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Psychiatrie - CHU de Strasbourg - France, Strasbourg, France